CLINICAL TRIAL: NCT06071338
Title: A Decision Support System Based on Classification Algorithms for the Diagnosis of Periodontal Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Abdulrahman Alshehri, Principal Investigator/Clinical Specialist, Ministry of Health, Saudi Arabia
Other Study IDs: H-06-B-091
Record Dates: First submitted 2023-09-22; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Periodontal Diseases
Keywords: periodontal; disease; diagnosis; machine; learning; Saudi
MeSH Terms: conditions — Periodontal Diseases; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Clinical Periodontal Examination — No details will be published from the clinical assessment.
  Other Names: orthopantomography Assessment

SUMMARY:
The study purposes For periodontal applications, such as diagnosing gingivitis and periodontal disease, artificial intelligence (AI) models have been developed; however, their accuracy and technological maturity are to be evolved. The applications of such technologies in the field of periodontics are walking baby steps worldwide. The Kingdom of Saudi Arabia is moving fast in technology adoption and implementation in different sectors. However, the healthcare sector, especially clinical-related, needs original research applied to Saudi subjects. The literature in the field of machine learning applications in dentistry is limited. Although AI models for periodontology applications are still being developed, they could serve as potent diagnostic instruments. The current study was planned to add to the current gap in the literature.

DETAILED DESCRIPTION:
A cross-sectional study design will be applied. Two hundred fifty patients will be evaluated by an experienced periodontist and used as input variables. The final diagnosis output will be generated by considering relevant information from the patient's medical history, clinical dental examination, and radiographic exam. Of the sample of 250 patients, 20% of the participants will be assigned randomly to the test group, while the rest will be assigned to the training group before feeding it to the algorithms.

The study purposes For periodontal applications, such as diagnosing gingivitis and periodontal disease, artificial intelligence (AI) models have been developed; however, their accuracy and technological maturity are to be evolved. The applications of such technologies in the field of periodontics are walking baby steps worldwide. The Kingdom of Saudi Arabia is moving fast in technology adoption and implementation in different sectors. However, the healthcare sector, especially clinical-related, needs original research applied to Saudi subjects. The literature in the field of machine learning applications in dentistry is limited. Although AI models for periodontology applications are still being developed, they could serve as potent diagnostic instruments. The current study was planned to add to the current gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or more
* no periodontal treatment has been done at least 6 months prior to the enrollment
* seeking periodontal treatment

Exclusion Criteria:

* refuse to volunteer in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be collected randomly during the study period planned to end by the end of the year 2023. Data will be collected from participants attending the periodontal department at Abha Specialized Dental Center seeking periodontal treatment.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Age | One time measure; baseline during periodontal clinical examination.
  <30, 30-34, 35-39, 40-44, 45-49, 50-54, 55-59, 60-64, 65-69, 70-74, 75-79, >80
Gender | One time measure; baseline during periodontal clinical examination.
  Male; Female.
Marital statue | One time measure; baseline during periodontal clinical examination.
  Married, widowed, divorced, never married
Education | One time measure; baseline during periodontal clinical examination.
  < secondary school, secondary school, graduate or equivalent, some college or associates degree, College graduate or higher
Physical Activities | One time measure; baseline during periodontal clinical examination.
  Light, Moderate, Heavy
Bleeding on Probing | One time measure; baseline during periodontal clinical examination.
  Yes; No
Gingival Index | One time measure; baseline during periodontal clinical examination.
  Percentage
Plaque Index | One time measure; baseline during periodontal clinical examination.
  Percentage
Periodontal Probing Depth | One time measure; baseline during periodontal clinical examination.
  PPD at the site of greatest loss (number)
Recession Type | One time measure; baseline during periodontal clinical examination.
  Yes; No
Clinical Attachment Loss | One time measure; baseline during periodontal clinical examination.
  CAL at the site of greatest loss (number)
Radiographic Bone Loss | One time measure; baseline during periodontal clinical examination.
  RBL at the site of greatest loss (percentage)
Tooth Mobility | One time measure; baseline during periodontal clinical examination.
  Yes; No
Missing Teeth | One time measure; baseline during periodontal clinical examination.
  Yes; No
Furcation Involvement | One time measure; baseline during periodontal clinical examination.
  Yes; No
Diabetes | One time measure; baseline during periodontal clinical examination.
  Healthy, <7% HbA1c,
  ≥7% HbA1c
Smoking | One time measure; baseline during periodontal clinical examination.
  None, <10 cig/day, ≥10cig/day
Body Mass Index | One time measure; baseline during periodontal clinical examination.
  Underweight, Healthy, Overweight, Obese
Cardiovascular Disease | One time measure; baseline during periodontal clinical examination.
  Yes; No

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman Al Shehri, BDS, MS, Principal Investigator — General Directorate of Health Affairs, Aseer Region, KSA.

IPD SHARING:
Plan to Share IPD: No
No intention and no need to share individual patient data with research community.

REFERENCES:
- [Result] Ozden FO, Ozgonenel O, Ozden B, Aydogdu A. Diagnosis of periodontal diseases using different classification algorithms: a preliminary study. Niger J Clin Pract. 2015 May-Jun;18(3):416-21. doi: 10.4103/1119-3077.151785. PMID 25772929
- [Result] Alqahtani HM, Koroukian SM, Stange K, Schiltz NK, Bissada NF. Identifying Factors Associated with Periodontal Disease Using Machine Learning. J Int Soc Prev Community Dent. 2022 Dec 30;12(6):612-622. doi: 10.4103/jispcd.JISPCD_188_22. eCollection 2022 Nov-Dec. PMID 36777017